CLINICAL TRIAL: NCT02552030
Title: iPhone App Compared to Standard RR-measurement - iPARR Trial
Brief Title: iPhone App Compared to Standard RR-measurement
Acronym: iPARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Eckstein (Other)
Collaborators: Preventicus GmbH (Industry)
Responsible Party: Sponsor-Investigator, Jens Eckstein, PD Dr. med, Leitender Arzt, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2015-287
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood pressure-measurement (Experimental): Seven repetitive blood pressure measurements will be performed the left or right arm of all participants with an iPhone 4s and a conventional oscillometric device 'cuff device (Omron HBP-1300-E Pro)'
  Interventions: Device: cuff device (Omron HBP-1300-E Pro); Device: iPhone 4s

INTERVENTIONS:
Device: cuff device (Omron HBP-1300-E Pro) — Comparison of systolic blood pressure results measured with an oscillometric cuff device (Omron HBP-1300-E Pro) and iPhone 4s
Device: iPhone 4s

SUMMARY:
In this Trial we compare a new application (App) running on an iPhone (Apple inc., Model 4S) to determine systolic blood pressure (RR) and compare it to conventional oscillometric measurements using an Omron HBP-1300-E Pro device. We will include 1000 participants and perform seven repetitive blood pressure measurements (3 iPhone, 4 Omron) in each person. Primary parameter will be the absolute difference (Delta) between the correlating blood pressure measurements in mmHg.

DETAILED DESCRIPTION:
Participants will be asked for consent at the University Hospital Basel at random based on availability. Recruitment is not limited to patients. After consenting patients will accompanied to a RR-measurement unit, positioned in a chair and kept at rest for 4 minutes. Then 7 blood pressure measurements at the same arm will be performed (Cuff/iPhone/Cuff/iPhone/Cuff/iPhone/Cuff). The Cuff measurement results will be documented in the source documents (mmHg) and transferred to a trial database. The iPhone data will be transferred with patient ID to "Preventicus" for calculation of the systolic blood pressure values (mmHg) based on the pulse waves recorded by transillumination of the index fingers of the participants. "Preventicus" will have NO access to the Cuff-measurement data. Then this data will be retransferred to the trial site and merged with help of the patient ID. Absolute and relative differences of the measured (Omron) and calculated (iPhone) systolic blood pressure values (mmHg) for will be calculated and published.

A subgroup of 40 participants will be evaluated in a highly standardized fashion according the ESH (European Society Hypertension) guidelines for validation studies. These data will then be published separately for validation purposes.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* in Sinus rhythm
* no anatomical limitation to take blood pressure

Exclusion Criteria:

* Atrial fibrillation
* Dialysis shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Absolute difference between systolic blood pressure values determined with an oscillometric cuff device and an iPhone 4s (Delta mmHg) | 1 day
  In each participant seven repetitive blood pressure measurements will be performed. Starting with a conventional cuff measurement followed by an iPhone measurement, followed by a conventional cuff measurement and so on. Then the absolute difference between each pair of successive measurements will be calculated. These differences will then be averaged and documented as primary result.

SECONDARY OUTCOMES:
Relative difference between oscillometric blood pressure measurement and iPhone based blood pressure measurement | 1 day
  Same as primary outcome, but calculation of delta (mmHg) and documentation as relative value (%) of the absolute systolic value.
Percent of invalid measurements | 1 day
  Percent of measurements that cannot be used for analysis
Comparison of primary outcome in the subgroup of patients with atherosclerosis compared to the participants without arteriosclerosis. | 1 day
  Quantitative differences between the accuracy of the iPhone measurements in the patients with known arteriosclerosis and the patients without arteriosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universityhospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorr M, Weber S, Birkemeyer R, Leonardi L, Winterhalder C, Raichle CJ, Brasier N, Burkard T, Eckstein J. iPhone App compared with standard blood pressure measurement -The iPARR trial. Am Heart J. 2021 Mar;233:102-108. doi: 10.1016/j.ahj.2020.12.003. Epub 2020 Dec 13. PMID 33321118
- [Derived] Vischer AS, Socrates T, Winterhalder C, Eckstein J, Mayr M, Burkard T. How should we measure blood pressure? Implications of the fourth blood pressure measurement in office blood pressure. J Clin Hypertens (Greenwich). 2021 Jan;23(1):35-43. doi: 10.1111/jch.14130. Epub 2020 Dec 14. PMID 33319471
- [Derived] Vischer AS, Mayr M, Socrates T, Winterhalder C, Leonardi L, Eckstein J, Burkard T. Impact of Single-Occasion American vs. Canadian Office Blood Pressure Measurement Recommendations on Blood Pressure Classification. Am J Hypertens. 2019 Jan 15;32(2):143-145. doi: 10.1093/ajh/hpy159. PMID 30371728
- [Derived] Raichle CJ, Eckstein J, Lapaire O, Leonardi L, Brasier N, Vischer AS, Burkard T. Performance of a Blood Pressure Smartphone App in Pregnant Women: The iPARR Trial (iPhone App Compared With Standard RR Measurement). Hypertension. 2018 Jun;71(6):1164-1169. doi: 10.1161/HYPERTENSIONAHA.117.10647. Epub 2018 Apr 9. PMID 29632098
- [Derived] Burkard T, Mayr M, Winterhalder C, Leonardi L, Eckstein J, Vischer AS. Reliability of single office blood pressure measurements. Heart. 2018 Jul;104(14):1173-1179. doi: 10.1136/heartjnl-2017-312523. Epub 2018 Mar 12. PMID 29530989
- See also: Developer of the tested App and responsible for blinded analysis of the iPhone data — http://www.preventicus.com